## **COVER PAGE**

**Title of document:** Randomized Controlled Study of Intraincisional Infiltration Versus Intraperitoneal Instillation of Standardized Dose of Ropivacaine 0.2% in Post-Laparoscopic Cholecystectomy Pain

NCT Number – Not Available

**Document Date** – 01/04/2014

**Informed Consent for Participation in Study** 

I agree to get myself/my patient to undergo laparoscopic cholecystectomy under GA at

Jawaharlal Nehru Medical College, Aligarh Muslim University, Aligarh. The effect and nature

of operation and anaesthesia and associated risks have been explained to me. I give consent

about the possible use of ropivacaine in my operation and fully understand that this is being

done in good faith and side-effects, if any, associated with its use, is part of treatment.

Signature of Patient:

Signature of Patient's Attendant:

Date of Consent:

Consent verified by (Name, Designation and Signature):